CLINICAL TRIAL: NCT06971978
Title: Pilot Randomized Controlled Trial To Assess the Effectiveness of a Heat Risk Reduction Decision Support Platform and Barriers and Facilitators of Its Implementation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Jeremy Hess, Professor: Environmental and Occupational Health Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00020944; 1P20ES036748-01 (NIH)
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Extreme Heat; Heat Health; Extreme Heat Waves; Heat; Emergency Preparedness; Disaster Management; Disaster Planning; Disasters
Keywords: heat; extreme heat event; climate; risk reduction
MeSH Terms: conditions — Risk Reduction Behavior | interventions — Hot Temperature; Risk Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive facilitated engagement with Chart. Chart is an online decision support platform designed to support evidence-based climate change adaptation. Chart has a risk assessment platform that provides estimates of heat-health risks at a census tract level under various hazard conditions. It also has a decision support platform that links drivers of risk in a given location with information about potential risk reduction activities and includes information useful to policymakers regarding intervention efficacy, timing, and cost. Facilitated engagement includes an initial introduction to the platform, real-time questions and answers, and focused discussion regarding priority interventions and planning and implementation needs. This engagement comprises about five hours of time that can be provided over the course of a couple weeks or several months, depending on the needs of the health department.
  Interventions: Other: Online decision support platform to support evidence-based heat health risk assessment and extreme heat event preparedness planning
- Control group (Active Comparator): Study participants in the control group will be provided with a package of information supportive of heat-health vulnerability and risk assessment and planning for risk reduction activities through built environment hazard mitigation and public health programming. This package will include an annotated list of online resources, including those available on Heat.gov and the CDC website, and a selected set of review papers on heat-health vulnerability, heat-health risk assessment, heat hazard mitigation through built environment strategies, and heat action planning and preparedness.
  Interventions: Other: Heat and health risk assessment and preparedness information

INTERVENTIONS:
Other: Online decision support platform to support evidence-based heat health risk assessment and extreme heat event preparedness planning — The intervention group will receive facilitated engagement with Chart. Chart is an online decision support platform designed to support evidence-based risk assessment and planning for extreme heat risk mitigation. Chart has a risk assessment platform that provides estimates of heat-health risks at a census tract level under various hazard conditions. It also has a decision support platform that links drivers of risk in a given location with information about potential risk reduction activities and includes information useful to policymakers regarding intervention efficacy, timing, and cost. Facilitated engagement includes an initial introduction to the platform, real-time questions and answers, and focused discussion regarding priority interventions and planning and implementation needs. This engagement comprises about five hours of time that can be provided over the course of a couple weeks or several months, depending on the needs of the health department.
  Arms: Intervention group
Other: Heat and health risk assessment and preparedness information — Study participants in the control group will be provided with a package of information supportive of heat-health vulnerability and risk assessment and planning for risk reduction activities through built environment hazard mitigation and public health programming. This package will include an annotated list of online resources, including those available on Heat.gov and the CDC website, and a selected set of review papers on heat-health vulnerability, heat-health risk assessment, heat hazard mitigation through built environment strategies, and heat action planning and preparedness.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if an innovative online decision support tool (Chart) that provides localized health risk assessment for extreme heat at the census tract level helps local health departments plan and prepare for extreme heat by identifying risk drivers in their jurisdictions, highlighting interventions that are effective for their jurisdiction's risk profile, and providing information regarding intervention implementation. This trial will evaluate barriers and facilitators of the tool's implementation. The main questions it aims to answer are:

1. Does a health department using the tool have better reach, effectiveness, adoption, implementation, and maintenance of heat-health activities compared with an information-only control?
2. What are the barriers and facilitators of Chart's implementation?

Researchers will compare health departments using Chart to health departments using provided heat-health information only.

ELIGIBILITY:
Inclusion Criteria:

* Local (city or county) health department
* Local (i.e., city or county) health department with at least partial autonomy to pursue the development and implementation of heat-health activities (i.e., not a state where all public health activities are administered at a state level)
* Availability of a staff member to participate in all elements of the trial. Local health department staff responsible for planning and implementing programming to protect constituents from extreme heat.
* Adults whose demographics and health status will mirror those of the general population.
* Current employees of included health departments aged 18 or greater

Exclusion Criteria:

* Being in a state where public health activities are exclusively managed at a state level and not having staff availability to participate
* Children and prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Baseline assessment: demographics | Baseline
  All departments will undertake the pre-intervention baseline assessment. The baseline assessment will gather information related to organizational demographics and demographics of the communities that the organization serves.
Baseline assessment: current activities | Baseline
  All departments will undertake the pre-intervention baseline assessment. The baseline assessment will gather information related to the organization's current activities relevant to extreme heat, including surveillance and program evaluation activities.
Baseline assessment: implementation factors | Baseline
  All departments will undertake the pre-intervention baseline assessment. The baseline assessment will gather information related to contextual and organizational factors that may affect intervention implementation.
Post-intervention survey: demographics | One year after the intervention begins.
  Meaningful changes in the demographics of the organization or service area.
Post-intervention survey: activities | One year after the intervention begins.
  The the post-intervention assessment will query participants regarding meaningful changes in the organization's activities and profile (e.g., the occurrence of a regional disaster that disrupted service provision across the organization).

SECONDARY OUTCOMES:
Key informant interviews | The key informant interviews will be completed one year after the intervention begins.
  Barriers and facilitators of Chart implementation and implementation outcomes using linkages to theoretical frameworks. Investigators will conduct key informant interviews (KIIs) with all 15 of the primary site contacts for the sites randomized to the intervention group. In this case, investigators will reference the Consolidated Framework for Implementation Research (CFIR) as a source of constructs to measure factors affecting Chart's implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Hess, MD, MPH, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hess J, Burden M, Isaksen TMB, Ebi KL, Errett NA, Gridley-Smith C, Kramer CB, McCarthy C, McLaughlin O, Patel R, Reed A, Smith MH, Wheat S, Sherr K. Pilot randomized controlled trial to assess the effectiveness of a heat risk reduction decision support platform and barriers and facilitators of its implementation. Implement Sci Commun. 2025 Nov 27;6(1):136. doi: 10.1186/s43058-025-00829-3. PMID 41310808